CLINICAL TRIAL: NCT05688839
Title: A Second Study to Assess the Efficacy and Safety of Jaktinib Hydrochloride Tablets in the Treatment of Severe Novel Coronavirus Pneumonia
Brief Title: A Study of Jaktinib Hydrochloride Tablets in the Treatment of Severe Novel Coronavirus Pneumonia
Acronym: COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK-IIT-005
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Novel COVID-19-Infected Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaktinib 100mg BID (Experimental): Jaktinib hydrochloride tablets, 2 x 50mg dosage, BID
  Interventions: Drug: Jaktinib hydrochloride tablets
- Placebo (Placebo Comparator): 2 x Placebo tablets, BID
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Jaktinib hydrochloride tablets — 2 doses per day, 100mg Jaktinib
  Arms: Jaktinib 100mg BID
Drug: placebo — 2 doses per day, placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo parallel control study and is expected to enroll 20-60 eligible patients with severe novel coronavirus pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old, regardless of gender;
* There is a history of novel coronavirus antigen- or nucleic acid-positive infection within 1-2 weeks;
* HRCT is consistent with the manifestation of viral pneumonia (judged by the investigator)
* Participants who voluntarily sign informed consent.

Exclusion Criteria:

* Participants who cannot take orally, or are suspected to be allergic to Jaktinib hydrochloride, similar drugs, or their excipients, or have severe gastrointestinal dysfunction that affects drug absorption;
* Critical pneumonia Participants with other organ failure requiring ICU monitoring and treatment;
* Participants who have received the following treatments within the specified time window before randomization:

  1. Participants have received Janus kinase (JAK) inhibitor, interleukin 6 (IL-6) inhibitor, IL-1 inhibitor, tumor necrosis factor (TNF) inhibitor, T cell or B cell depletion agent, interferon and other immunosuppressive drugs within the first two weeks of randomization, except glucocorticoid;
  2. Systematically used CYP 3A4 potent inhibitor or potent inducer in the first five drug half-lives at random;
* Immune deficiency;
* Participants who have received the novel coronavirus vaccine within 1 week before randomization;
* Prior to randomization, there were the following active and uncontrolled infections: tuberculosis, HIV, syphilis, mycoplasma, chlamydia, parasites, and viral infections other than SARS CoV-2 that required systemic anti-infection treatment;
* Renal diseases requiring dialysis treatment;
* Pregnant and lactating women;
* Any other Participants that were considered unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects with disease progression or all-cause mortality
Efficacy of Jaktinib | 14 days after randomization
  The proportion of subjects with disease progression or all-cause mortality
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects whose (National Institute of Allergy and Infectious Disease Ordinal Scale (NIAID-OS) score improved by ≥ 2 points from the baseline
Efficacy of Jaktinib | 28 days after randomization
  The change value of NIAID-OS score compared with the baseline
Efficacy of Jaktinib | Up to 28 days after randomization
  Time interval from randomization to clinical improvement (defined as NIAID-OS 1-3 points)
Efficacy of Jaktinib | Up to 28 days after randomization
  Time interval from randomization to discharge
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects receiving mechanical ventilation due to disease progression at 3, 7, and 14 days after randomization until the end of treatment (EOT)
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects whose chest High-Resolution CT (HRCT) showed significant absorption of pulmonary inflammation (definition of significant absorption: the lung inflammatory lesions were reduced by more than 50%) at 7, 14 days after treatment until EOT

SECONDARY OUTCOMES:
Safety of Jaktinib | Up to 2 months after randomization
  Incidence rate of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: RongHu Li, Principal Investigator — Changsha Taihe Hospital
Locations (1):
- Changsha Taihe Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No